CLINICAL TRIAL: NCT05865977
Title: Diaphragmatic Tissue Doppler Imaging During a Spontaneous Breathing Trial to Predict Extubation Failure in Preterm Infants
Brief Title: dTDI During a SBT to Predict Extubation Failure in Preterm Infants
Status: Recruiting | Type: Observational
Sponsor: Wang Jianhui (Other)
Responsible Party: Sponsor-Investigator, Wang Jianhui, Attending doctor, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: 20230223
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Premature
Keywords: tissue Doppler imaging; Premature infants; extubation; diaphragm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the failure group: Re-intubation within 48 h after passing the SBT was defined as failed weaning.
  Interventions: Device: diaphragmatic tissue Doppler imaging，dTDI
- the success group: Extubation and invasive mechanical ventilation was not needed within 48 h after extubation was defined as successful weaning.
  Interventions: Device: diaphragmatic tissue Doppler imaging，dTDI

INTERVENTIONS:
Device: diaphragmatic tissue Doppler imaging，dTDI — dTDI was performed at the end of the SBT to assess excursion, velocity, and acceleration.

SUMMARY:
Weaning from mechanical ventilation is a critical issue and the diaphragmatic disfunction has been demonstrated to play an important role in extubation failure. the aim of present investigation is to evaluate diaphragmatic excursion velocity during in patients undergoing spontaneous breathing trial through tissue Doppler analysis in both inspiration and expiration.

ELIGIBILITY:
Inclusion Criteria:

* premature infants with gestational age <32 weeks and supported by invasive mechanical ventilation ≥48 hours
* All the indications for extubation are met：cough or vomiting due to spontaneous breathing and sputum aspiration; ventilator parameters in recent 24 hours: MAP < 8cmH2O, RR < 30 times/min, FiO2 < 30%; Arterial blood gas: pH > 7.25, (PaCO2< 60mmHg, BE < 8mmol/L, oxygen saturation > 90%
* a successful SBT
* parents or legal guardians sign informed consent to attend this study

Exclusion Criteria:

* accidental extubation
* chest CT or bronchoscopy during hospitalization indicated congenital airway dysplasia
* complex congenital heart disease
* congenital metabolic diseases, neuromuscular diseases
* severe brain injury
* surgical mechanical ventilation
* give up before extubation;
* pneumothorax or pleural effusion
* no consent is signed

Ages: 2 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: premature infants with gestational age <32 weeks and supported by invasive mechanical ventilation ≥48 hours
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-25 (Actual); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Change in diaphragmatic displacement velocity | an average of 20 minutes
  Inspiratory and expiratory diaphragmatic displacement velocity evaluated with tissue doppler during the assisted ventilation modality which preceded the trial, during the spontaneous breathing trial and in spontaneous breathing.

SECONDARY OUTCOMES:
Diaphragmatic acceleration and deceleration | an average of 20 minutes
  Diaphragmatic acceleration and deceleration evaluated with tissue doppler during the assisted ventilation modality which preceded the trial, during the spontaneous breathing trial and in spontaneous breathing.
Gas exchange - arterial carbon dioxide tension | through each trial completion, an average of 20 minutes
  Arterial blood gases sample
Gas exchange - pH | an average of 20 minutes
  Arterial blood gases sample
Gas exchange - arterial oxygen tension | an average of 20 min
  Arterial blood gases sample
Silverman Andersen Respiratory Severity Score (SA-RSS) | an average of 20 min
  SA-RSS to assess work of breathing after extubation.
Number of patients who experienced weaning failure | 48 hours
  the need for non invasive ventilation or re-intubation due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China